CLINICAL TRIAL: NCT00100555
Title: A Study of the Clinical Safety, Tolerability, and Efficacy of Zoledronic Acid Compared to an Oral Bisphosphonate
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CZOL446H2315
Record Dates: First submitted 2005-01-03; First posted 2005-01-04 (Estimated); Last update posted 2012-04-27 (Estimated); Status verified 2012-04

CONDITIONS: Osteoporosis
Keywords: Osteoporosis, osteopenia, post-menopausal, zoledronic acid
MeSH Terms: conditions — Osteoporosis; Bone Diseases, Metabolic | interventions — Zoledronic Acid

INTERVENTIONS:
Drug: zoledronic acid

SUMMARY:
The purpose of this trial is to study the clinical safety, tolerability, and efficacy of zoledronic acid compared to an oral bisphosphonate in postmenopausal women with osteoporosis.

ELIGIBILITY:
Inclusion Criteria:

* Postmenopausal women between 45 and 79 years of age
* Must be osteopenic/osteoporotic

Exclusion Criteria:

* Any women of child-bearing potential

Other protocol-defined inclusion/exclusion criteria may apply.

Ages: 45 Years to 79 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120
Dates: Start 2004-06; Primary Completion 2005-06 (Actual); Study Completion 2005-06 (Actual)

PRIMARY OUTCOMES:
Assess the rapidity of onset of action on bone turnover by comparing the percent change from baseline in urine N-telopeptide (NTx) in post-menopausal women

SECONDARY OUTCOMES:
To assess the effect on markers of bone turnover by comparing the percent change from baseline in serum C-telopeptide (CTx) and urine NTx in post-menopausal women
To assess the frequency, intensity, and "bothersomeness" of dyspepsia, as measured by the Nepean Dyspepsia Index - Short Form, Symptom Checklist
To assess patient preferences for annual i.v. therapy compared to weekly oral therapy

CONTACTS AND LOCATIONS:
Locations (18):
- United States (18):
  - Univ. of Alabama/Division of Clinical Immunology and Rheumatology, Birmingham, Alabama
  - Radiant Research, San Diego, California
  - Denver Arthritis Clinic, Denver, Colorado
  - Florida Medical Research Institute, Gainesville, Florida
  - Northwestern Center for Clinical Research, Chicago, Illinois
  - The Center for Rheumatology and Bone Research, Wheaton, Maryland
  - Midwest Arthritis Center, Kalamazoo, Michigan
  - St. John's Medical Research, Springfield, Missouri
  - Deaconess Billings Clinic Research Division, Billings, Montana
  - UMDNJ-Robert Wood Johnson Medical School, New Brunswick, New Jersey
  - Helen Hayes Hospital - Regional Bone Clinic, West Haverstraw, New York
  - Private Practice, Mayfield Village, Ohio
  - The Arthritis Clinic of Jackson, Jackson, Tennessee
  - Radiant Research, Dallas, Texas
  - Univ. of North Texas Health Science Center at Fort Worth, Fort Worth, Texas
  - St. Luke's Episcopal Hospital Ctr for Ortho. Res. and Education, Houston, Texas
  - Women's Health Center, Salt Lake City, Utah
  - Valley Medical Associates, Lewisburg, West Virginia